CLINICAL TRIAL: NCT07086209
Title: Optimizing Hamstring Rehabilitation With Amino Acids: A Randomized Controlled Study for Seamless Return to Sports in Football Athletes
Brief Title: Optimizing Hamstring Rehabilitation With Amino Acids
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Kamal Hadib Abdulridha, PhD Student, Universidad de Zaragoza
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: Unizar
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Seamless Return to Sports
Keywords: Hamstring Rehabilitation; Return to play; Amino Acids; Football
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic Exercise + Amino Acid Supplementation (Experimental): Participants in this arm will undergo a structured 6-week therapeutic exercise rehabilitation program combined with daily oral branched-chain amino acid (BCAA) supplementation (10 g per day, divided into two doses: pre-training and post-training). The exercise program includes progressive isometric, eccentric, plyometric, and sprint-specific training to optimize hamstring recovery.
  Interventions: Dietary Supplement: Branched-Chain Amino Acid Supplement; Behavioral: Therapeutic Exercise Program
- Therapeutic Exercise Only (Active Comparator): Arm Description:
  Participants in this arm will undergo the same structured 6-week therapeutic exercise rehabilitation program without any amino acid supplementation. The exercise program includes progressive isometric, eccentric, plyometric, and sprint-specific training for hamstring recovery.
  Interventions: Dietary Supplement: Branched-Chain Amino Acid Supplement; Behavioral: Therapeutic Exercise Program

INTERVENTIONS:
Dietary Supplement: Branched-Chain Amino Acid Supplement — Oral BCAA blend (leucine, isoleucine, valine), 10 g/day divided into two doses, pre- and post-training, for 6 weeks.
  Other Names: Therapeutic Exercise + Amino Acid Supplementation
Behavioral: Therapeutic Exercise Program — 6-week structured program including isometric, eccentric, plyometric, and sprint-specific exercises.

SUMMARY:
Hamstring injuries are among the most prevalent and troublesome injuries in athletes, particularly those engaged in sports that require high-speed movements such as sprinting, kicking, and rapid changes in direction. The hamstring muscles, which include the biceps femoris, semitendinosus, and semimembranosus, are essential for powerful lower limb actions, and thus, any injury to these muscles can significantly impact an athlete's performance and recovery. These injuries often occur during eccentric muscle contractions, such as when the muscles lengthen rapidly under tension, as seen in running and sprinting. According to epidemiological studies, hamstring strains account for a substantial portion of sports-related injuries, with hamstring strains being the most commonly reported injury in disciplines such as football, soccer, rugby, and athletics. In professional football, for instance, hamstring injuries account for approximately 12% of all injuries and represent the most frequent muscle strain, underlining their significance in the context of athletic performance.

ELIGIBILITY:
Inclusion Criteria:

* • Male football players aged 18 to 35 years.

  * Active players from eight clubs in the Iraqi Football League.
  * MRI-confirmed partial hamstring muscle injury.
  * No participation in other ongoing rehabilitation programs.

Exclusion Criteria:

* • History of hamstring injury in the past six months.

  * Any other musculoskeletal injuries affecting lower limbs.
  * Contraindications for MRI scanning (e.g., metal implants, pacemakers).
  * Any existing neurological or metabolic conditions affecting muscle recovery.

Max Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-09-19 (Estimated); Primary Completion 2025-10-19 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Change in Hamstring Muscle Strength | Baseline, Mid-Rehabilitation (Week 3), Post-Rehabilitation (Week 6)
  Isometric knee flexion strength measured at 15° and 90° using the ForHealth Kit to assess change from baseline.

SECONDARY OUTCOMES:
MRI Findings | Baseline and Post-Rehabilitation (Week 6)
  MRI assessment of muscle healing, including reduction in edema and tear resolution.

OTHER OUTCOMES:
Adherence to Rehabilitation | Throughout 6-week intervention period
  Percentage of rehabilitation sessions attended by each participant, tracked via attendance logs.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: pubmed — https://pubmed.ncbi.nlm.nih.gov/